CLINICAL TRIAL: NCT06058598
Title: High Intensity Interval Training in Patients With Glaucoma
Brief Title: Exercise Training in Patients With Glaucoma
Acronym: HIT GLAUCOMA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henner Hanssen (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other); University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor-Investigator, Henner Hanssen, Professor, University of Basel
Organization: University of Basel (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-01397
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-07

CONDITIONS: Glaucoma, Open-Angle; Exercise Training; Microvascular Health
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Exercise

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Group performing exercise training and receiving standard care
  Interventions: Other: Exercise Training
- Control Group (Experimental): Group receiving lifestyle counseling and receiving standard care
  Interventions: Other: Lifestyle Counselling

INTERVENTIONS:
Other: Exercise Training — 6-months supervised exercise training + 6 months unsupervised exercise training
  Arms: Intervention Group
Other: Lifestyle Counselling — 12-months of lifestyle counselling
  Arms: Control Group

SUMMARY:
HIT GLAUCOMA is a multicenter exercise study for glaucoma patients between three institutes: the Department of Sport, Exercise and Health (DSBG) of the University of Basel, the Eye Clinic at the University Hospital Basel and the UZ Leuven (Belgium). The main objective of the study is to investigate the possibility of using exercise therapy to treat glaucoma. Participants will be randomly divided into two groups: Intervention and Control group. The intervention group will receive a high-intensity interval training plan, and the control group will receive lifestyle counseling and standard therapy. With this method, the study aims to validate an exercise therapy concept that could significantly improve disease progression and quality of life in patients with glaucoma.

DETAILED DESCRIPTION:
Approximately 57.5 million people are affected by primary open-angle glaucoma, and it is estimated that this number will increase to 111.8 million by 2040. Despite the high prevalence and critical outlook of the disease, the pathogenesis of glaucoma is still not fully understood and treatment options remain inadequate. In particular, for glaucoma with normal intraocular pressure, there is as yet no evidence-based effective treatment option. This particular type of glaucoma may, in part, be the result of impaired microvascular endothelial function. Physical training has a proven effect on vascular health; because glaucoma involves a vascular component, positive effects of high-intensity interval training can be assumed. Thus, it could be an effective treatment for glaucoma disease.

Patients will be randomly assigned to either the intervention or control group. Patients assigned to the intervention group will participate in a 6-month exercise training program followed by a 6-months non-supervised and home-based physical activity maintenance program. During the first 6 months, patients in the intervention group participate in 18 supervised exercise sessions at the DSBG, interspersed by unsupervised exercise interventions at home.

All patients will be seen at baseline, after three months and six months of aerobic exercise training, and after another six months of physical activity and exercise self-maintenance (intervention group) or control condition. Each subject will be asked to undergo standard ophthalmic examination, non-invasive retinal assessments, peripheral blood withdrawal, and additional peripheral vascular examinations. The study design is based on regular glaucoma follow-up intervals (every 6 months) and does not intervene with clinical care and governmental reimbursement of standard care. Patients will finish their study participation after 6 months of exercise training followed by 6 months of physical activity and exercise self-maintenance or control condition.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent of the participant has been obtained prior to any screening procedures
* Patients with primary open angle glaucoma (POAG), high tension glaucoma (HTG) and normal tension glaucoma (NTG), aged 40 - 75 years
* In regular follow-up in either of the two study centres

Exclusion Criteria:

* Patients having had glaucoma surgery within 6 months before start of the project
* Patients with changes in topical medication or laser trabeculoplasty within 3 months before start of the project
* Patients with very severe glaucoma (visual field mean deviation lower than -12Db)
* Significant opacification of ocular media
* Patients with life-threatening arrhythmia, signs of ischemia during CPET which preclude participation in an exercise trial
* Patients with insulin treated diabetes, chronic obstructive pulmonary disease or cancer.
* Patients doing ≥1 structured exercise training session per week or >150min of exercise/week assessed via the following two questions: a. On average, how many days per week do you engage in moderate to vigorous physical activity (like brisk walking)? b. On average, how many minutes per day do you engage in physical activity at this level? Calculate the total weekly minutes of exercise by multiplying a times b.
* Mental or physical limitation precluding participation in a high intensity exercise program

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Microvascular health: retinal arteriolar and venular dilation and diameters | 6-months
  Retinal arteriolar and venular flicker light-induced dilation after six months; Retinal arteriolar and venular diameters after six months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Basel, Department of Sport, Exercise & Health, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Van Eijgen J, Schuhmann V, Fingerroos EL, Renier M, Burchert H, Kropfl JM, Van Craenenbroeck A, Cornelissen V, Gugleta K, Stalmans I, Hanssen H. High-intensity interval training in patients with glaucoma (HIT-GLAUCOMA): protocol for a multicenter randomized controlled exercise trial. Front Physiol. 2024 May 16;15:1349313. doi: 10.3389/fphys.2024.1349313. eCollection 2024. PMID 38818519